CLINICAL TRIAL: NCT01504646
Title: Randomized Controlled Trial of Marine Lipid Fraction PCSO-524™ on Airway Inflammation and Hyperpnea-Induced Bronchoconstriction in Asthma
Brief Title: Effect of a Component of Fish Oil on Exercise-Induced Bronchoconstriction and Airway Inflammation in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Pharmalink (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1108006502
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2013-04

CONDITIONS: Asthma; Exercise-Induced Bronchoconstriction
Keywords: Asthma; Exercise-Induced Bronchoconstriction; lipids; n-3 PUFA; airway inflammation; Bronchoconstriction
MeSH Terms: conditions — Asthma | interventions — lyprinol; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olive Oil Capsule (Placebo Comparator): Ten subjects will take eight placebo olive oil capsules per day for three weeks.
  Interventions: Dietary Supplement: Placebo (Olive Oil)
- Lyprinol (Experimental): Ten subjects will take eight Lyprinol capsules per day for three weeks.
  Interventions: Dietary Supplement: Lyprinol

INTERVENTIONS:
Dietary Supplement: Lyprinol — 8 capsules (1 capsule=50mg n-PUFA, 100mg olive oil) per day for 3 weeks
  Arms: Lyprinol
Dietary Supplement: Placebo (Olive Oil) — 8 capsules (1 capsule = 100mg olive oil) per day for 3 weeks
  Other Names: Olive Oil
  Arms: Olive Oil Capsule

SUMMARY:
The primary aim of this study will be to evaluate the effects of Lyprinol® supplementation on airway inflammation and the bronchoconstrictor response to dry air hyperpnea in individuals with asthma. The investigators hypothesize that Lyprinol® supplementation, compared to placebo, will significantly attenuate airway inflammation and hyperpnea-induced bronchoconstriction in asthmatic individuals.

DETAILED DESCRIPTION:
Our research group has shown, on numerous occasions that fish oil has a markedly protective effect in suppressing airway inflammation and exercise-induced bronchoconstriction in elite athletes and asthmatic individuals. Purified fish oil and the marine lipid fraction PCSO-524™ (Lyprinol™) have both been used in supplementation studies in asthma [2, 10, 11]. While fish oil is a rich source of the omega-3 fatty acids eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), Lyprinol® is a patented extract of stabilized lipids from the New Zealand green-lipped mussel, Perna canaliculus, combined with olive oil and vitamin E. EPA and DHA are the main ingredients of fish oil, and thus there will be similarities between Lyprinol and fish oil in terms of mechanism of action. Thus, we are aiming to show that Lyprinol® can modulate these inflammatory eicosanoids to exert anti-inflammatory effects.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with asthma and EIB. Evidence of a diagnosis of asthma will include medication use as well as history and symptoms as outlined in the NHLBI Guidelines for the Diagnosis and Management of Asthma. For the diagnosis of EIB, subjects must demonstrate a fall in FEV1 of ≥ 10% after dry air eucapnic voluntary hyperventilation (EVH), a simulated exercise challenge; FEV1 is a measure of lung function
* Not currently be taking any fish oil supplements
* Limit their fish consumption to 1 fish meal per week during the course of the study

Exclusion Criteria:

* Severe asthma is indicated. These subjects will be identified by a post-EVH drop in FEV1 that is greater than 50% during their first lab testing session or will have a history of severe asthma-related events such as hospitalizations or emergency room visits. Only mild to moderate asthmatics (i.e. subjects whose FEV1 drops by 10-50%) will be included in this study.
* They taking currently taking asthma maintenance medications
* They are pregnant
* They have a history of hyperlipidemia (high cholesterol), hypertension, diabetes, bleeding disorder, delayed clotting time, or seizure disorder
* They are allergic to shellfish, fish, corn, or soy products

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function (Percent Change in FEV1, measured in Liters) | 8 weeks
  The percent change in FEV1 is the percent change in the volume of air exhaled during the first second of a forced exhalation as measured before and after the surrogate exercise challenge.

SECONDARY OUTCOMES:
Fraction of Exhaled Nitric Oxide | 8 weeks
  The concentration of exhaled Nitric Oxide (measured as parts per billion) will be measured using a Nitric Oxide Analyzer.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Health, Physical Education, and Recreation, Bloomington, Indiana, United States

REFERENCES:
- [Background] Crapo RO, Casaburi R, Coates AL, Enright PL, Hankinson JL, Irvin CG, MacIntyre NR, McKay RT, Wanger JS, Anderson SD, Cockcroft DW, Fish JE, Sterk PJ. Guidelines for methacholine and exercise challenge testing-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. Am J Respir Crit Care Med. 2000 Jan;161(1):309-29. doi: 10.1164/ajrccm.161.1.ats11-99. No abstract available. PMID 10619836
- [Background] Mickleborough TD. A nutritional approach to managing exercise-induced asthma. Exerc Sport Sci Rev. 2008 Jul;36(3):135-44. doi: 10.1097/JES.0b013e31817be827. PMID 18580294
- [Background] Dahlen B, Roquet A, Inman MD, Karlsson O, Naya I, Anstren G, O'Byrne PM, Dahlen SE. Influence of zafirlukast and loratadine on exercise-induced bronchoconstriction. J Allergy Clin Immunol. 2002 May;109(5):789-93. doi: 10.1067/mai.2002.123306. PMID 11994701
- [Background] Horrocks LA, Yeo YK. Health benefits of docosahexaenoic acid (DHA). Pharmacol Res. 1999 Sep;40(3):211-25. doi: 10.1006/phrs.1999.0495. PMID 10479465
- [Background] Flower RJ, Perretti M. Controlling inflammation: a fat chance? J Exp Med. 2005 Mar 7;201(5):671-4. doi: 10.1084/jem.20050222. PMID 15753201
- [Background] Soutar A, Seaton A, Brown K. Bronchial reactivity and dietary antioxidants. Thorax. 1997 Feb;52(2):166-70. doi: 10.1136/thx.52.2.166. PMID 9059479
- [Background] Mickleborough TD, Lindley MR, Ionescu AA, Fly AD. Protective effect of fish oil supplementation on exercise-induced bronchoconstriction in asthma. Chest. 2006 Jan;129(1):39-49. doi: 10.1378/chest.129.1.39. PMID 16424411
- [Background] Mickleborough TD, Murray RL, Ionescu AA, Lindley MR. Fish oil supplementation reduces severity of exercise-induced bronchoconstriction in elite athletes. Am J Respir Crit Care Med. 2003 Nov 15;168(10):1181-9. doi: 10.1164/rccm.200303-373OC. Epub 2003 Aug 6. PMID 12904324